CLINICAL TRIAL: NCT00804375
Title: Study of the Efficacy, Safety and Tolerability of Topical 2PX (Strontium Chloride Hexahydrate) in Patients With Chronic, Moderate-to-severe Lower Limb Post-amputation Stump Pain.
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Smerud Medical Research International AS (Other)
Collaborators: SantoSolve AS (Industry)
Responsible Party: Thorfinn Ege, SantoSolve AS
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2PX-SP-02; SMR-1850
Record Dates: First submitted 2008-12-05; First posted 2008-12-08 (Estimated); Last update posted 2010-03-24 (Estimated); Status verified 2010-03

CONDITIONS: Stump Pain
Keywords: stump pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 2PX (Experimental): Pain medication
  Interventions: Drug: 2PX
- placebo (Placebo Comparator): placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: 2PX — cutaneous solution to be applied twice daily for 84 days
  Arms: 2PX
Drug: Placebo — cutaneous solution to be applied twice daily for 84 days
  Arms: placebo

SUMMARY:
Primary: To compare the analgesic effect over 12 weeks of topical 2PX in stump pain.

Secondary: To prospectively measure other efficacy and safety variables of topical 2PX in stump pain. Exploratory analyses will be performed to measure efficacy and safety variables of topical 2PX in phantom pain

ELIGIBILITY:
Inclusion Criteria:

* Lower limb amputation at least 6 months prior to Visit 1. Amputation must be transtibial, transfemoral or through the knee. For patients with transfemoral amputation, the point of amputation must be ≥10 cm from the inguinal region.
* Presenting with moderate-to-severe stump pain. For the purpose of this study, the following criteria must all apply:

  1. Stump pain commencing post amputation and continues at Visit 1 despite continued use of analgesic medication
  2. Stump pain present on a daily basis
  3. Stump pain intensity as Average stump Pain Intensity (AsPI) ≥40 on 100 mm VAS at Screening
  4. Stump pain intensity at the randomisation visit: Mean (over the 7 day run-in period) AsPI rating ≥40 on a 100 mm VAS.
  5. Pain at the site of the extremity amputation. The pain is located mainly in the stump itself. (Patients with concurrent phantom pain may be enrolled in the study.)
  6. Stump pain persists despite proper healing of the stump
* Outpatients, aged 18 years and above
* Underlying therapy (e.g., rehabilitation procedures, analgesia, physio-therapy, spinal cord stimulation (except for topical or subcutaneous local analgesics)) may be continued throughout the duration of the study, if the regimen has been stable during the 4 weeks immediately prior to Visit 1. If underlying therapy is continued during the study the regimen must be maintained for the duration of the study.
* Written informed consent

Exclusion Criteria:

* Patients with forefoot amputations alone are excluded from participation.
* Patients who have received treatment with any topical or subcutaneously administered analgesic agent for stump or phantom pain in the 4 weeks prior to study entry (i.e. Visit 1).
* Underlying therapy (e.g., rehabilitation procedures, analgesia, physio-therapy, spinal cord stimulation) is not permitted if the regimen has not been stable in the 4 weeks immediately prior to Visit 1.
* After the 7 day run-in phase: patients taking any new or changing the dose of any underlying analgesic medication (except for rescue medication as defined in this protocol).
* Patients with open wounds, burns or other non-intact skin at site(s) of study drug administration (unhealed stumps).
* Patients with significant discomfort from their prosthesis limiting use of the prosthesis. Use of a prosthesis is not a requirement for participation in the study.
* Pregnancy
* Female patients of childbearing potential unwilling to use adequate contraception measures throughout the duration of the study. For the purpose of this study, adequate contraception is defined as:

  * oral, injected or implanted hormonal methods of contraception; OR
  * placement of an intrauterine device (IUD) or intrauterine system (IUS); OR
  * barrier methods of contraception: Condom or occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/suppository Note: Male sterilization or abstinence are not acceptable methods of birth control and would preclude enrolment in the study.

Note: For post-menopausal women: less than 12 months since the last spontaneous menstrual bleeding will exclude the patient unless they are willing to utilise acceptable methods of contraception for the duration of the study.

* Breast-feeding/lactating mothers
* Any active malignant disease (except basal cell carcinoma; BCC)
* Patients who have previously received 2PX.
* Patients requiring concomitant administration of strontium ranelate (Protelos®)
* Patients who have received an investigational drug or used an investigational device within the 30 days prior to study entry.
* Patients unable to comply with the study assessments
* Patients with documented or suspected current alcohol or drug abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2008-12; Primary Completion 2010-06 (Estimated); Study Completion 2010-06 (Estimated)

PRIMARY OUTCOMES:
Average (stump) Pain Intensity (AsPI): and recorded in the diary in response to the question: 'What was your average stump pain intensity over the past 24 hours?' on a 100 mm VAS (0 = no pain, 100 = worst pain imaginable). | will be measured each evening (at least 1 hour after taking off the prosthesis, if applicable, and immediately prior to administering the evening dose of study medication)

SECONDARY OUTCOMES:
Worst (stump) Pain Intensity (WsPI): recorded in the diary in response to the question: 'What was your worst stump pain level during the past 24 hours?' on a 100 mm VAS (0 = no pain, 100 = worst pain imaginable). | will be measured each evening (at least 1 hour after taking off the prosthesis, if applicable, and immediately prior to administering the evening dose of study medication

CONTACTS AND LOCATIONS:
Overall Officials: Lone Nikolajsen, MD, Principal Investigator — Aarhus University Hospital
Locations (19):
- Denmark (3):
  - Site in Århus, Aarhus
  - Site in Herlev, Herlev
  - Site in Hvidovre, Hvidovre
- Site in Wiesbaden, Wiesbaden, Germany
- Norway (4):
  - Site in Ålesund, Ålesund
  - Site in Hamar, Hamar
  - Site in Oslo, Oslo
  - Site in Stavern, Stavern
- Russia (2):
  - Site in St. Petersburg, Saint Petersburg
  - Site in St.Petersburg, Saint Petersburg
- United Kingdom (9):
  - Site in Belfast, Belfast
  - Site in Birmingham, Birmingham
  - Site in Edinburgh, Edinburgh
  - Site in Glasgow, Glasgow
  - Site in Hammersmith, Hammersmith
  - Site in Crystal Palace, London
  - Site in Manchester, Manchester
  - Site in Middlesborough, Middlesbrough
  - Site in Newcastle, Newcastle